CLINICAL TRIAL: NCT05803200
Title: Maternal and Infant Characteristics and Outcomes Following Exposure to HyQvia During Pregnancy: A Case Series Study Based on US Claims Data
Brief Title: A Study to Describe Mothers' and Babies' Outcomes After Exposure to HyQvia During Pregnancy
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-771-4004; EUPAS103800 (Other: The European Union electronic Register of Post-Authorisation Studies (EU PAS Register))
Record Dates: First submitted 2023-03-14; First posted 2023-04-07 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Exposure During Pregnancy
Keywords: Drug Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HyQvia: Pregnant female participants who have insurance coverage with full prescriptions benefits exposed to HyQvia during the period from 90 days before the last menstrual period (LMP) through 30 days after delivery will be observed retrospectively from 1 January 2014 to 31 December 2020 (up to 7 years).
  Interventions: Drug: No intervention

INTERVENTIONS:
Drug: No intervention — No intervention was given as this is an observational study.

SUMMARY:
The main aim of this study is to provide further information on the safety profile of HyQvia during pregnancy. This will be done by checking the characteristics of the mother and their babies. They will also be checked for any safety outcomes that will occur when exposed to HyQvia during pregnancy.

DETAILED DESCRIPTION:
This is a non-interventional, retrospective, case series of commercially insured pregnant women exposed to HyQvia during their pregnancy identified according to the MarketScan Research Database. This study will assess maternal characteristics, patterns of HyQvia utilization and pregnancy outcomes in all pregnancies exposed to HyQvia during pregnancy.

This study will enroll approximately at least 7 patients based on feasibility assessment. Participants will be enrolled in the following cohort:

• HyQvia

This study will have a retrospective data collection from 1 January 2014 to 31 December 2020. This study would be conducted in the US.

The overall time for data collection in this study will be approximately 7 years.

ELIGIBILITY:
Inclusion criteria • Exposed to HyQvia in the etiologic window defined as 90 days prior to the LMP until the end of pregnancy.

Exclusion criteria

• NA

Ages: 16 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Pregnant females who were exposed to HyQVia during pregnancy would be enrolled in the study.
Study Population: Commercially insured US pregnant women exposed to HyQvia from 90 days before LMP to the end of pregnancy and their infants included in the MarketScan Research Database during the period 2014-2020.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-04-14 (Actual); Study Completion 2023-04-14 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Major Congenital Malformations in the Infant | Up to 7 years
  A major malformation is defined as a structural abnormality with surgical, medical, or cosmetic importance. Data for infants will be reviewed in the database from the date of delivery to 90 days following birth to check for any malformations. The number of infants with malformations during the database period of 1 January 2014 to 31 December 2020 (up to 7 years) will be reported.
Number of Participants with Spontaneous Abortion | Up to 7 years
  Spontaneous abortion is defined as pregnancy loss before 20 weeks of gestation.
Number of Participants with Stillbirth | Up to 7 years
  Stillbirth is defined as a fetal death after 20 weeks of gestation.
Number of Participants with Preterm Birth | Up to 7 years
  Pre-term birth is defined as delivery before 37 weeks of gestation.
Number of Participants Being Small for Gestational Age (SGA) | Up to 7 years
  SGA will be defined as weight at birth of full and preterm live-born infants in <10th percentile.
Number of Participants with Admission to Neonatal Intensive Care Unit (NICU) | Up to 7 years
  NICU admissions will be identified by current procedure terminology (CPT) codes in maternal and infant claims within 30 days of delivery.
Number of Participants With Any Major Clinical Diagnosis or Procedures | Up to 7 years
  Major clinical diagnoses include preeclampsia, post-partum hemorrhage, infections and thrombosis while procedures include cesarean section.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/e25fff0d9a404d43?idFilter=%5B%22TAK-771-4004%22%5D